CLINICAL TRIAL: NCT04710823
Title: Ultrasound- Guided Continuous Serratus Anterior Plane Block Versus Ultrasound- Guided Continuous Thoracic Paravertebral Block For Analgesia in Multiple Traumatic Rib Fractures.
Brief Title: Ultrasound- Guided Continuous Serratus Anterior Plane Block Versus Ultrasound- Guided Continuous Thoracic Paravertebral Block in Multiple Traumatic Rib Fractures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Rehab, Principal Investigator; Assistant lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32596/09/18
Record Dates: First submitted 2021-01-11; First posted 2021-01-15 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Serratus Anterior Plane Block; Thoracic Paravertebral Block; Ultrasound; Multiple Traumatic Rib Fractures; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic paravertebral block (Experimental): Patients will receive ultrasound-guided continuous thoracic paravertebral blockusing bupivacaine 0.25% for 4 days.
  Interventions: Procedure: Thoracic paravertebral block
- Serratus anterior plane block (Experimental): Patients will receive ultrasound-guided continuous SAP block using bupivacaine 0.25% for 4 days.
  Interventions: Procedure: Serratus anterior plane block

INTERVENTIONS:
Procedure: Thoracic paravertebral block — A bolus dose of 0.25% bupivacaine (0.3 ml/kg) will be injected slowly over 3-5 minutes. At 30 minutes after injection of the loading dose, the dermatomal loss of sensation to pinprick was tested. Patients who reported pain to pinprick will be considered to have a failed block and were excluded from the study. The block will be maintained by continuous infusion of bupivacaine 0.25% at a rate of 0.1 ml/kg/h via a syringe pump. The infusion will be continued for 4 days.
  Arms: Thoracic paravertebral block
Procedure: Serratus anterior plane block — A bolus of 30 ml of 0.25% bupivacaine will be injected slowly over 3-5 minutes between latissmus dorsi muscle and serratus anterior muscle (Figure 15). Then a catheter was inserted through the Tuohy needle and advanced 3cm into the space and secured in place. At 30 minutes after injection of a loading dose, the dermatomal loss of sensation to pinprick will be tested. Patients who reported pain to pinprick will be considered to have a failed block and were excluded from the study. The block will be maintained by continuous infusion of bupivacaine 0.25% at a rate of 0.1 ml/kg/h via a syringe pump. The infusion was continued for 4 days.
  Arms: Serratus anterior plane block

SUMMARY:
The aim of this study is to compare the analgesic efficacy of ultrasound guided continuous SAP block and ultrasound guided continuous TPVB in patients with multiple traumatic rib fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender aged between 22-65 years with unilateral traumatic multiple fracture ribs (≥ 3 fractured ribs).

Exclusion Criteria:

* • Contraindications to regional block such as patient's refusal, coagulopathy, local infection at the site of the block, known allergy to local anesthetic drugs and spinal deformity.

  * Patients suffer from severe cardiovascular disease, hepatic or renal disease and patients with history of psychiatric illness.
  * Patients had indications for mechanical ventilation on admission or during the study period.
  * Patients had indications for immediate surgery for other associated injuries.
  * Patients with hemodynamic instability.
  * Patients having spine or pelvic fracture, traumatic brain injury, altered conscious level or spinal cord injury.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Degree of pain scores | Four days after the block
  Pain will be assessed at rest and on coughing using the VAS on a scale from 0 (no pain) to 100 (worst pain) before the block, 30 minutes, 60 minutes after the block, and then every six hours for 4 days. But in order not to interrupt the sleeping pattern of patients, patients will be considered pain free (VAS= 0) if they will be at sleep with no tachypnea, tachycardia, or hypertension.

SECONDARY OUTCOMES:
Total consumption of morphine | Four days after the block
  Rescue analgesia will be provided with morphine (0.05 mg/kg) intravenously if visual analogue score (VAS) ≥ 40.
Changes of forced vital capacity (FVC) | Four days after the block
  Forced vital capacity (FVC) will be assessed using bedside spirometry before the block, 30 minutes, 60 minutes after the blocks, and then every eight hours for 4 days
Changes of forced expiratory volume in one second (FEV1) | Four days after the block
  Forced expiratory volume in one second (FEV1) will be assessed using bedside spirometry before the block, 30 minutes, 60 minutes after the blocks, and then every eight hours for 4 days
Changes of forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) | Four days after the block
  FEV1/FVC ratio will be assessed using bedside spirometry before the block, 30 minutes, 60 minutes after the blocks, and then every eight hours for 4 days
Length of ICU stay | Four days after the block
  Length of ICU stay, defined as the time from admission to ICU to time of transfer to the surgical ward.
Length of hospital stay | Four days after the block
Incidence of complications | Four days after the block
  Incidence of respiratory complications and mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon a reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: After 3 months from the end of study and for one year